CLINICAL TRIAL: NCT07370194
Title: Investigating the Impact of Serum Potassium Levels on Prevalence and Risk Factors Associated With Management Strategies for Patients With Hyperkalaemia in Brazilian Clinical Settings: An Observational Study.
Brief Title: Observational Study on the Prevalence and Risk Factors of Patients With Hyperkalaemia in Brazil
Acronym: HOPE
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9480R00075
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hyperkalemia
Keywords: serum potassium levels
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a descriptive, retrospective study involving patients from private cardiology, nephrology, and dialysis clinics in Brazil who participated in the National Hyperkalaemia Diagnosis Campaign. The study used anonymised data from the Hi Technologies Ltda. database. The objective was to estimate and characterise the prevalence of hyperkalaemia (HK), as well as to analyse the demographic profile, clinical characteristics, risk factors and treatment patterns associated with total blood potassium levels.

DETAILED DESCRIPTION:
The aim of this study is to describe the clinical and demographic profile, as well as the prevalence of hyperkalaemia and its associated risk factors in patients who participated in the First National Campaign for the Diagnosis of Hyperkalaemia through the incorporation of a point-of-care device, with potassium results available during the consultation. The data used in this study consists of anonymised records. The study population will consist of adults aged 18 years or older, of both sexes, with a medical history of heart failure, diabetes mellitus, chronic kidney disease, and/or systemic arterial hypertension, who attended cardiology, nephrology, or dialysis clinics between April and November 2025.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older; Pre-existing comorbidities, including: o Heart failure (regardless of phenotype); o Chronic kidney disease (any stage); o Diabetes mellitus; o Systemic arterial hypertension.

Exclusion Criteria:

* Diagnosis of advanced malignant neoplasm undergoing palliative treatment; Other advanced diseases with a life expectancy of less than one year; Patients with no information on risk factors for hyperkalaemia (HK).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adults aged 18 years or older, of both sexes, with a medical history of heart failure, diabetes mellitus, chronic kidney disease, and/or systemic arterial hypertension, who attended cardiology, nephrology, or dialysis clinics between April and November 2025.
Sampling Method: Probability Sample
Enrollment: 6215 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Hyperkalemia | through study completion, an average of 1 year
  To provide a comprehensive characterisation of the prevalence of hyperkalaemia in patients with high-risk comorbidities treated at private cardiology, nephrology, and dialysis clinics in Brazil.
Epidemiological and Clinical Characterisation | through study completion, an average of 1 year
  Identify clinical, demographic, and therapeutic factors associated with serum potassium levels.

SECONDARY OUTCOMES:
Practical and Social Impact | through study completion, an average of 1 year
  Expand knowledge about the clinical profile of patients with HK, supporting the development of screening, prevention, and early management strategies for a safer and more personalised approach.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/